CLINICAL TRIAL: NCT00010036
Title: A Phase I/II Trial of CPT-11 With Carboplatin in Patients With Glioblastoma Multiforme Prior to Radiation Therapy
Brief Title: Carboplatin Plus Irinotecan in Treating Patients With Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068435; P30CA016087 (NIH); NYU-9902; P-UPJOHN-986475197; NCI-G00-1909
Record Dates: First submitted 2001-02-02; First posted 2003-09-04 (Estimated); Last update posted 2011-03-28 (Estimated); Status verified 2011-03

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma | interventions — Carboplatin; Irinotecan; Radiotherapy

INTERVENTIONS:
Drug: carboplatin
Drug: irinotecan hydrochloride
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining carboplatin with irinotecan in treating patients who have glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose (MTD) of carboplatin and irinotecan in patients with glioblastoma multiforme. (Phase I closed to accrual as of 6/24/02)
* Determine the toxic effects of this regimen in these patients.
* Determine the objective response in patients treated with the established MTD of this regimen.
* Determine time to tumor progression and survival of patients treated with this regimen.

OUTLINE: This is a dose-escalation study. Patients in the phase II portion of the study are stratified according to age (under 60 vs 60 and over), ECOG performance status (0-1 vs 2), and extent of resection (total vs subtotal). (Phase I closed to accrual as of 6/24/02)

Within 4 weeks of surgery, patients receive carboplatin IV over 30 minutes followed by irinotecan IV over 90 minutes on day 1. Treatment repeats every 4 weeks for a maximum of 6 courses in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of carboplatin and irinotecan until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. Once the MTD is determined, additional patients are accrued to receive carboplatin and irinotecan at the recommended phase II dose. (Phase I closed to accrual as of 6/24/02)

After chemotherapy, all patients undergo radiotherapy.

Patients are followed for 30 days.

PROJECTED ACCRUAL: A total of 24-107 patients (3-54 for phase I and 21-53 for phase II) will be accrued for this study. (Phase I closed to accrual as of 6/24/02)

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed glioblastoma multiforme
* Measurable disease
* No CNS metastases or carcinomatous meningitis

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2 OR
* Karnofsky 70-100%

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Granulocyte count greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3
* Hemoglobin at least 9.0 g/dL

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* SGOT no greater than 3 times upper limit of normal (ULN) (5 times ULN if liver involvement)
* No known Gilbert's syndrome

Renal:

* Creatinine no greater than 1.5 mg/dL

Cardiovascular:

* No myocardial infarction within the past 6 months
* No congestive heart failure requiring therapy

Other:

* HIV negative
* No active or uncontrolled infection
* No psychiatric disorder that would preclude study
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer or carcinoma in situ of the cervix
* No uncontrolled diabetes mellitus (i.e., random blood sugar of 200 mg or more)
* No other severe disease that would preclude study
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior immunotherapy or biologic therapy
* No concurrent sargramostim (GM-CSF)
* No concurrent filgrastim (G-CSF) with course 1
* No concurrent immunotherapy

Chemotherapy:

* No prior chemotherapy
* No other concurrent chemotherapy

Endocrine therapy:

* Must have maintained a stable or decreasing dose of corticosteroids for 2 weeks prior to study
* Concurrent corticosteroids for cerebral edema allowed
* No concurrent anticancer hormonal therapy

Radiotherapy:

* No prior radiotherapy
* No concurrent radiotherapy

Surgery:

* At least 2 weeks since prior surgery

Other:

* No other concurrent investigational agent or participation on any other clinical study
* No concurrent immunosuppressive drugs
* No concurrent phenobarbital or valproic acid
* No concurrent anticonvulsants except carbamazepine or gabapentin
* No concurrent prochlorperazine on day of irinotecan treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1999-05; Primary Completion 2001-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael L. Gruber, MD, Study Chair — NYU Langone Health
Locations (1):
- NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York, United States